CLINICAL TRIAL: NCT01396642
Title: Effect of Topical Emollient Therapy on Clinical Outcomes in Preterm Neonates - A Clinical Trial
Brief Title: Topical Emollient Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Principal Investigator, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1258-CHS/ERC-09
Record Dates: First submitted 2011-07-07; First posted 2011-07-19 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Blood Stream Infection
Keywords: Topical Emollient Therapy; Emollient; Preterm; Hospital Acquired Infection
MeSH Terms: conditions — Premature Birth; Cross Infection | interventions — Emollients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical Emollient (Experimental): Neonates in this group will receive topical emollient application with coconut oil twice a day till 28th day of life
  Interventions: Other: Topical Emollient
- Routine Skin Care (No Intervention): Neonates in this group will receive routine skin care as per unit protocol

INTERVENTIONS:
Other: Topical Emollient — Neonates in this group will receive topical emollient application with coconut oil twice a day till 28th day of life
  Arms: Topical Emollient

SUMMARY:
Almost all (99%) of the neonatal deaths occur in lower and middle income countries. Most of these deaths are attributable to prematurity and infection. With the increasing rate of premature births in some settings, the mortality rate of over 50% among preterm babies in some of the developing countries require inexpensive hospital-based strategies to prevent fatal infections in newborns of these countries. As most of the deaths in preterm neonates are attributable to their vulnerability of infection, a potential low cost intervention like topical emollient therapy can be effectively directed to reduce infection related mortality and morbidity in the developing countries. Topical emollient therapy reduces the rate of infection by enhancing the skin barrier function, thus reducing trans-epidermal water loss consequently conserving heat and energy to promote growth.

The broad goal of the study is to improve the survival rate of hospitalized preterm neonates in the developing countries by decreasing the incidence of infection using low-cost interventions.

HYPOTHESIS:

It is hypothesized that topical emollient therapy with coconut oil twice a day till 28th day of life in hospitalized preterm neonates reduces the incidence proportion of hospital acquired infection by 40% 15 as compared to routine skin care. For the secondary objective it is hypothesized that the weight gain in the neonates receiving prophylactic application of emollient, which is coconut oil twice a day till 28th day of life, is at least 2g/kg/day18 more as compared to the weight gain in the routine skin care group.

DETAILED DESCRIPTION:
Research question:

1. The primary research question to be addressed via this study is whether the prophylactic application of emollient, which is coconut oil twice a day till 28th day of life, effective in reducing the incidence proportion of hospital acquired infection among preterm neonates by 40% as compared to the routine skin care.
2. The secondary research question is whether the weight gain in the neonates receiving prophylactic application of emollient, which is coconut oil twice a day till 28th day of life, is at least 2g/kg/day more as compared to the weight gain in the routine skin care group.

Objectives: This study has the following primary objectives:

1. To evaluate the effectiveness of topical emollient in preventing hospital acquired infection in preterm neonates.

   The secondary objective is:
2. To compare the weight gain among the two groups of neonates.

ELIGIBILITY:
Inclusion Criteria:

1. Any preterm neonates (>26 weeks and < 37 weeks of gestation by maternal dates)
2. Birth weight of at least 750 gm
3. Age ≤72 hours of life
4. Baseline blood cultures obtained
5. Expected survival > 48 hours (based on the clinical judgment by the physicians)

Exclusion Criteria:

1. Neonate with severe RDS on admission as declared by the consulting Physician on the basis of radiologic findings.
2. Neonate within first 24 hours of critical care
3. Life threatening congenital anomalies
4. Congenital skin anomalies
5. Hydrops Fetalis
6. Congenital infection of the skin
7. History of any previous treatment with the ointment
8. Newborns admitted for major surgical procedure with expected high rates of infectious complications.
9. Newborns with positive baseline blood cultures

Ages: 5 Minutes to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 258 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Hospital Acquired Blood Stream Infection | 28 days of life
  Hospital Acquired Infection is defined as a blood culture positive for any organism in a neonate with baseline negative cultures on admission.

SECONDARY OUTCOMES:
Weight Gain | 28th Day of Life

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar ZB Bhutta, MBBS, PhD, Principal Investigator — Aga Khan University; Rehana A Salam, MSc, Principal Investigator — Aga Khan University
Locations (1):
- The Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Salam RA, Darmstadt GL, Bhutta ZA. Effect of emollient therapy on clinical outcomes in preterm neonates in Pakistan: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2015 May;100(3):F210-5. doi: 10.1136/archdischild-2014-307157. Epub 2015 Jan 30. PMID 25637007